CLINICAL TRIAL: NCT02035930
Title: Effect of Dexmedetomidine on Bispectral Index and Propofol Requirements During Different Menstrual Cycle
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Geng guiqi, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: TWang
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Abnormal Menstrual Cycle
Keywords: Bispectral Index Monitor, Menstrual Cycle, Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- menstrual cycle,dexmedetomidine (Other)
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine

SUMMARY:
The study was done to evaluate the effects of the follicular and luteal phases of the menstrual cycle on sedation level at loss of consciousness and bispectral index reach to 50 during propofol anesthesia, in patients with and without preoperative intravenous dexmedetomidine .

ELIGIBILITY:
Inclusion Criteria:

* a regular menstrual cycle
* elective gynecologic surgery

Exclusion Criteria:

* pregnancy
* breastfeeding
* obesity
* known hypersensitivity to drugs used in the study protocol;
* use of psychotropic drugs and steroids within 72 hours before the surgery
* central nervous system injury
* renal impairment
* alcoholism and opioid addiction.

Ages: 24 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
bispectral index at loss of eyelash reflex | up to 2 years

SECONDARY OUTCOMES:
propofol requirements from propofol administered to loss of eyelash reflex and bispectral index reduced to 50 | up to 2 years

OTHER OUTCOMES:
duration from propofol administered to loss of eyelash reflex and bispectral index reduced to 50 | up to 2 years